CLINICAL TRIAL: NCT01346800
Title: Pharmacokinetic Interaction Between Ritonavir and Prasugrel in Healthy Volunteers
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: University Hospital, Geneva (Other)
Responsible Party: Pr Jules Desmeules, University Hospitals, Geneva
Allocation: Non-Randomized | Model: Crossover | Masking: None | Purpose: Basic Science
Other Study IDs: MICRO-PRASU-RITONAVIR
Record Dates: First submitted 2011-04-21; First posted 2011-05-03 (Estimated); Last update posted 2011-10-06 (Estimated); Status verified 2011-04

CONDITIONS: Healthy Volunteers
MeSH Terms: interventions — Prasugrel Hydrochloride; Ritonavir

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Prasugrel 10mg po (Experimental)
  Interventions: Drug: Prasugrel
- Prasugrel 10mg po + ritonavir 100mg po (Experimental)
  Interventions: Drug: Prasugrel; Drug: Ritonavir

INTERVENTIONS:
Drug: Prasugrel — Assessment of prasugrel metabolic ratio and phenotyping of CYP2B6/2C9/2C19/3A4
Drug: Ritonavir — Assessment of prasugrel metabolic ratio and phenotyping of CYP2B6/2C9/2C19/3A4 in presence of ritonavir
  Arms: Prasugrel 10mg po + ritonavir 100mg po

SUMMARY:
HIV patients are at particular risk to develop cardiovascular disease (CVD) as they exhibit multiple known risk factors for CVD. Of specific concern is the fact that use of the non nucleosidic reverse transcriptase inhibitors (NNRTI) and/or protease inhibitors (PI) drug classes is associated with dyslipidemia known to increase the risk of coronary heart disease particularly among older subjects with normalized CD4 cell counts and suppressed HIV replication. HIV patients could thus potentially receive anti-aggregant therapy concomitantly with their antiretroviral treatment. Prasugrel is an anti-aggregating agent indicated to prevent the recurrence of ischemic events after coronary arteries stenting. It is a pro-drug mainly metabolized by cytochromes P450 (CYP) 3A and 2B6 and to a lesser extent by CYP2C9 and 2C19. Ritonavir is an anti-protease and CYP3A4 and CYP2B6 inhibitor used in anti-HIV therapy. The aim of the present study is to assess the potential drug-drug interaction between prasugrel and the CYP3A/2B6 inhibitor ritonavir. Ten healthy volunteers will receive prasugrel 10mg alone or after 100mg ritonavir. The effect of ritonavir on prasugrel pharmacokinetics will be assessed. The two sessions will be separated by a one-week "wash out" period. During each session, CYP3A, 2B6, 2C9 and 2C19 activities will be assessed by a micrococktail approach with microdoses of midazolam, bupropion, flurbiprofen and omeprazole. The pharmacokinetics of prasugrel active metabolite will be assessed during the two sessions.

ELIGIBILITY:
Inclusion Criteria:

* Healthy male volunteers aged from 18 to 60 years
* BMI between 18 and 25
* Understanding of French language and able to give an inform consent.

Exclusion Criteria:

* smoker
* hypersensitivity to prasugrel or ritonavir or constituents of the tablets - - regular alcohol consumption
* concomitant disease
* intake of any drug or particular food (grapefruit) that can affect or metabolized by the CYP3A, 2C19, 2B6 and 2C9 within 1 month before the study
* pathologies or drugs associated with an increased bleeding risk such as aspirin, non-steroidal anti-inflammatory drugs, steroids and serotonin reuptake inhibitors (in the last 10 days before the start of the study)
* bleeding familial history or antecedent or haemorrhagic disease
* previous gastro-intestinal ulcer or active ulcer

Ages: 18 Years to 60 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 10 (Actual)
Dates: Start 2011-02; Primary Completion 2011-06 (Actual); Study Completion 2011-09 (Actual)

PRIMARY OUTCOMES:
Plasmatic prasugrel metabolites concentrations (ng/mL) in presence/absence of ritonavir | One week
  The concentrations will be measured at 9 differents times during 6 hours (0,1min,30min,1H,1H30,2H,3H,4H,6H). The measurements will be repeated one week later for 6 hours

SECONDARY OUTCOMES:
CYP2B6 phenotype in presence/absence of ritonavir | One week
  The phenotype will be assessed by taking a blood sample once and one week later
CYP2C9 phenotype in presence/absence of ritonavir | one week
  The phenotype will be assessed by taking a blood sample once and one week later
CYP2C19 phenotype in presence/absence of ritonavir | one week
  The phenotype will be assessed by taking a blood sample once and one week later
CYP3A4 phenotype in presence/absence of ritonavir | one week
  The phenotype will be assessed by taking a blood sample once and one week later

CONTACTS AND LOCATIONS:
Overall Officials: Jules A Desmeules, Pr, Principal Investigator — University Hospital, Geneva
Locations (1):
- University Hospitals, Geneva, Switzerland